CLINICAL TRIAL: NCT05818748
Title: Effect Of Virtual Reality Distraction on Symptom Control and Anxiety in Children With Leukemia: A Randomized Controlled Trial
Brief Title: Effect Of Virtual Reality Distraction on Symptom Control and Anxiety in Children With Leukemia
Acronym: VR-Ege
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dokuz Eylul University (Other)
Collaborators: Ege University (Other)
Responsible Party: Principal Investigator, Gülçin Özalp Gerçeker, pHD, Assoc. Prof., Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: VR Ege
Record Dates: First submitted 2023-03-30; First posted 2023-04-19 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Symptom Cluster; Anxiety
MeSH Terms: conditions — Syndrome; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomised
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- virtual reality distraction (Experimental): watching the application by wearing virtual glasses to the child during the 1st, 2nd and 3rd days of chemotherapy treatment
  Interventions: Device: virtual reality
- control (No Intervention): no virtual reality distraction

INTERVENTIONS:
Device: virtual reality — virtual reality distraction
  Arms: virtual reality distraction

SUMMARY:
This study aim to evaluate the effect of virtual reality distraction on symptom management and anxiety in children aged 7-18 years with leukemia.

DETAILED DESCRIPTION:
While the virtual reality initiative was applied to the children in the study group, no harm was given to the children in the control group. The virtual reality distraction method will not be applied to the control group. After the child and his family are informed about the study, their written informed consent will be obtained.

When the patients were admitted to the clinic the day before chemotherapy treatment was started, the symptom screening scale and anxiety scale will be applied.

Control Group: The researcher stated that no additional procedure will be applied to the children in the control group and that the symptom screening scale and anxiety measurement will be obtained by explaining that he/she should evaluate the scale every day for 3 days.

VR group; A distraction intervention will be applied for 10-15 minutes once a day with VR glasses. The symptom screening scale and anxiety measurement will be obtained by explaining that he/she should evaluate the scale every day for 3 days.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients aged 7-18 years receiving leukemia treatment in the Pediatric Hematology Service
* 4 weeks after diagnosis (not in the induction phase)
* No need for blood product transfusion (less than 8 mg/dl for hematological malignancies, less than 7 mg/dl for oncological malignancies)
* Consent to voluntarily participate in the study and written consent from the child and parent

Exclusion Criteria:

* The child has a physical and psychological deficit that will prevent him from wearing glasses to watch virtual reality
* Having a symptom of nausea and vomiting
* Being in a terminal period
* Undergoing a surgical operation
* Unwillingness to participate in the study
* Having a history of vertigo (having a history of train, motion sickness)
* The child and family do not know Turkish

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-03-30 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Change in symptom cluster | during the 1st, 2nd and 3rd days of chemotherapy treatment
  Symptom by Symptom Screening Tool(8-18) in SSPedi-Pediatric Patients with Cancer
Change in anxiety | (during the 1st, 2nd and 3rd days of chemotherapy treatment)
  anxiety by State-Trait Anxiety Inventory for Children

CONTACTS AND LOCATIONS:
Overall Officials: Gülçin Özalp Gerçeker, pHD, Study Director — Dokuz Eylul University
Locations (2):
- Turkey (Türkiye) (2):
  - Gülçin Özalp Gerçeker, Izmir
  - Figen Yardımcı, Izmir

IPD SHARING:
Plan to Share IPD: No